CLINICAL TRIAL: NCT06947759
Title: Application of 18F-FDG PET/MRI as an Initial Staging Procedure for Locally Advanced Nasopharyngeal Carcinoma
Brief Title: Application of 18F-FDG PET/MRI for Initial Staging in Locally Advanced Nasopharyngeal Carcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CF25181A; TCVGH-1142401F (Other Grant/Funding Number: Taichung Veterans General Hospital)
Record Dates: First submitted 2025-04-17; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-03

CONDITIONS: Nuclear Medicine; Oncology
Keywords: PET/MRI; Nasopharyngeal carcinoma; EBV DNA
MeSH Terms: conditions — Neoplasms; Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Radiation: PET/MRI — This single-center prospective observational study targets patients pathologically diagnosed with nasopharyngeal carcinoma (NPC) and clinically staged as cT3-4/N2-N3. Participants will first undergo standard whole-body 18F-FDG PET/CT, followed by localized 18F-FDG PET/MRI of the head and neck within 4 hours. Both imaging procedures will be performed according to standard clinical protocols to ensure data consistency and comparability.
  PET/MRI data will be independently interpreted by an experienced nuclear medicine physician and a radiologist. The sensitivity, specificity, and staging accuracy for detecting distant metastases will be analyzed. In cases of disagreement, a third physician will mediate to reach a consensus.
  The study team will also record the operational time, direct costs, and potential issues encountered during the examination process for both imaging modalities. All participants will be followed for at least one year to validate imaging results and assess correlation

SUMMARY:
This single-center prospective observational study aims to evaluate the feasibility, cost-effectiveness, and clinical value of positron emission tomography/magnetic resonance imaging (PET/MRI) for initial staging in patients with locally advanced nasopharyngeal carcinoma (NPC). It will compare the diagnostic performance of PET/MRI, including sensitivity, specificity, and staging accuracy, with traditional staging methods such as positron emission tomography/computed tomography (PET/CT).

Nasopharyngeal carcinoma is prevalent in Southeast Asia and North Africa, with approximately 5% of newly diagnosed cases presenting with distant metastases. For patients with N2-3 disease and elevated Epstein-Barr virus (EBV) DNA levels, the risk of distant metastasis can reach 27.5%. Accurate detection of distant metastases at diagnosis is crucial for staging and treatment planning. Current National Comprehensive Cancer Network (NCCN) guidelines recommend fluorodeoxyglucose (18F-FDG) PET/CT for staging in locally advanced nasopharyngeal carcinoma, as traditional tools (e.g., chest CT, abdominal ultrasound, bone scans) may yield false-negative results.

PET/MRI, as a novel imaging technique, offers potential advantages such as improved diagnostic accuracy, shorter scan times, and reduced false-positive rates. However, its clinical application is limited by high costs and equipment availability. This study will explore the clinical value and economic feasibility of PET/MRI in nasopharyngeal carcinoma staging, aiming to establish its potential role in improving diagnostic pathways.

DETAILED DESCRIPTION:
1. Background:

   Nasopharyngeal carcinoma (NPC) is prevalent in Southeast Asia and North Africa, with 5% of newly diagnosed cases showing distant metastases. For N2-3 stage patients with high Epstein-Barr virus (EBV) DNA levels, the metastasis rate can reach 27.5%. Accurate detection at diagnosis is crucial for staging and treatment planning. While the National Comprehensive Cancer Network (NCCN) recommends fluorodeoxyglucose (18F-FDG) positron emission tomography/computed tomography (PET/CT) for staging locally advanced NPC, traditional methods like chest CT or ultrasound may yield false negatives. PET/MRI offers improved accuracy and reduced false positives but is limited by high costs and low accessibility. This study examines the cost-effectiveness and clinical value of PET/MRI in NPC staging.
2. Material and methods:

   This study is a single-center prospective observational study. It will recruit patients aged 18 years or older with pathologically confirmed nasopharyngeal carcinoma (NPC) who have not received any NPC-related treatment and agree to participate. All participants will undergo PET/CT and PET/MRI to compare their diagnostic performance in detecting distant metastases, including sensitivity, specificity, and staging accuracy. The study will also evaluate the time efficiency and cost-effectiveness of PET/MRI to explore its clinical value and limitations.
3. Expecting Results:

This study aims to demonstrate that PET/MRI has superior diagnostic accuracy over PET/CT in staging locally advanced nasopharyngeal carcinoma, especially in detecting distant metastases. Despite higher costs, PET/MRI's accuracy may streamline diagnosis, reduce unnecessary tests, and support precise treatment strategies, improving patient outcomes and quality of life. The results will provide evidence for its clinical use and guide future diagnostic improvements.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically diagnosed with nasopharyngeal carcinoma (NPC) through endoscopic biopsy at the hospital's otolaryngology department.
* Clinically staged as cT3-4/N2-N3.
* Age: 18 years and older.
* Participants must voluntarily sign an informed consent form, acknowledging understanding of the study objectives and potential risks.

Exclusion Criteria:

* Patients with poorly controlled diabetes. -Patients with a history of head and neck malignancies or a history of non- head and neck cancers with no evidence of disease for at least 3 years.
* Patients with clinical staging of cT1-2N0-1.
* Patients with factors that may affect PET/MRI image quality, such as implanted metal devices or MRI contraindications, or those with a history of contrast agent allergies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants in this study are pathologically diagnosed nasopharyngeal carcinoma (NPC) patients, primarily focusing on those with locally advanced staging (cT3-4/N2-N3), who have not yet received any treatment related to NPC. Participants must be 18 years or older, in good physical condition, and able to cooperate in completing imaging examinations and treatments.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of PET/MRI vs. PET/CT in Detecting Distant Metastases in NPC | 1 year
  This study evaluates the sensitivity of PET/MRI compared to PET/CT in detecting distant metastases in nasopharyngeal carcinoma (NPC). Sensitivity is analyzed to determine the ability of each modality to accurately identify true-positive cases, validated through pathological confirmation and follow-up data.
Specificity Comparison Between PET/MRI and PET/CT in Detecting Distant Metastases in NPC | 1year
  This study evaluates the specificity of PET/MRI and PET/CT in detecting distant metastases in nasopharyngeal carcinoma (NPC). Specificity, defined as the ability to correctly identify true-negative cases, is validated using pathological confirmation and follow-up data to assess the diagnostic accuracy of each imaging modality.
Comparison of Overall Accuracy Between PET/MRI and PET/CT in Detecting Distant Metastases in NPC | 1 year
  This study compares the overall accuracy of PET/MRI and PET/CT in detecting distant metastases in nasopharyngeal carcinoma (NPC). Overall accuracy is defined as the proportion of correct results (both true positives and true negatives) among all the cases, validated by pathological confirmation and follow-up data to assess the diagnostic effectiveness of each imaging modality.

SECONDARY OUTCOMES:
Comparison of Examination Costs Between PET/MRI and PET/CT in NPC Staging | 1 year
  This study compares the examination costs of PET/MRI and PET/CT in staging nasopharyngeal carcinoma (NPC). The analysis includes the direct costs associated with each imaging modality, such as equipment, personnel, and operational expenses, to evaluate the cost-effectiveness of both techniques in clinical practice.

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

REFERENCES:
- [Background] Feng Q, Liang J, Wang L, Ge X, Ding Z, Wu H. A diagnosis model in nasopharyngeal carcinoma based on PET/MRI radiomics and semiquantitative parameters. BMC Med Imaging. 2022 Aug 29;22(1):150. doi: 10.1186/s12880-022-00883-6. PMID 36038819
- [Background] Fang Y, Chen S, Xu Y, Qiang M, Tao C, Huang S, Wang L, Chen X, Cao C. Assessment of bone lesions with 18 F-FDG PET/MRI in patients with nasopharyngeal carcinoma. Nucl Med Commun. 2023 Jun 1;44(6):457-462. doi: 10.1097/MNM.0000000000001682. Epub 2023 Mar 10. PMID 36897049
- [Background] Cao C, Fang Y, Yu B, Xu Y, Qiang M, Tao C, Huang S, Chen X. Use of 18F-FDG PET/MRI as an Initial Staging Procedure for Nasopharyngeal Carcinoma. J Magn Reson Imaging. 2024 Mar;59(3):922-928. doi: 10.1002/jmri.28842. Epub 2023 May 31. PMID 37256732